CLINICAL TRIAL: NCT00643656
Title: Study of the Efficiency of Kalinox 170 Bar During Liver Biospy of Focal Lesion
Brief Title: Use of 50% Nitrous Oxide / 50% Oxygen Premix During Liver Biopsy of Focal Lesion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT : 2006-004203-19
Record Dates: First submitted 2008-03-19; First posted 2008-03-26 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Liver Biopsy
Keywords: Liver biopsy
MeSH Terms: interventions — Oxygen; Nitrogen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Mixture of 50% nitrous oxide and 50% oxygen
  Interventions: Drug: Kalinox 170 bar
- B (Placebo Comparator): Mixture of 50% oxygen and 50% nitrogen
  Interventions: Drug: Mix of 50% oxygen and 50% nitrogen

INTERVENTIONS:
Drug: Kalinox 170 bar — Flow of gas administrated to the patient between 4 and 15 litre/min and less than 1 hour
  Arms: A
Drug: Mix of 50% oxygen and 50% nitrogen — Flow of gas administrated to the patient between 4 and 15 litre/min and less than 1 hour
  Arms: B

SUMMARY:
A 50% nitrous oxide / 50% oxygen premix is administrated to the patient during the realization of liver biopsy in order to relax him and to reduce his pain during this painful medical treatment. This single investigator centre and national clinical trial is done blindly : half of patients will receive 50% nitrous oxide / 50% oxygen premix and half of them a placebo gas (mixture of 50% oxygen and 50% nitrogen). 94 patients will be included in this clinical protocol.

ELIGIBILITY:
Inclusion Criteria:

* patient requiring a liver biopsy of focal lesion
* Age upper than 18 years
* OMS : 0 to 3
* patient consent form signed

Exclusion Criteria:

* patient unable to use Visual Analog Scale (VAS)
* OMS upper than 3
* coagulation disorder
* contraindication linked to the experimental product
* patient already included in another clinical trial uncompatible with this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain measurement by using Visual Analog Scale (VAS) | At the end of the liver biospy

SECONDARY OUTCOMES:
Patient's acceptance and doctor's satisfaction | At the end of the liver biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- Beaujon hospital, Clichy, France

REFERENCES:
- [Background] Meskine N, Vullierme MP, Zappa M, d'Assignies G, Sibert A, Vilgrain V. Evaluation of analgesic effect of equimolar mixture of oxygen and nitrous oxide inhalation during percutaneous biopsy of focal liver lesions: a double-blind randomized study. Acad Radiol. 2011 Jul;18(7):816-21. doi: 10.1016/j.acra.2011.01.025. Epub 2011 Apr 20. PMID 21511500
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/21511500/